CLINICAL TRIAL: NCT05456984
Title: The PsychOsis and Diabetes Service Model (PODS) Population Profile Study.
Status: Completed | Type: Observational
Sponsor: King's College London (Other)
Collaborators: Burdett Trust for Nursing (Other)
Responsible Party: Sponsor
Other Study IDs: 307600
Record Dates: First submitted 2022-03-25; First posted 2022-07-13 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Type2Diabetes; Severe Mental Disorder
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
People with severe mental illness (SMI), defined as psychotic and bipolar disorders, die 17-20 years earlier than the general population, the most common cause of death being cardiovascular diseases (CVD). The major contributor to CVD mortality in SMI is the increased prevalence of type 2 diabetes (T2D) compared to the general population. T2D is a paradigm of a single condition that progresses to multiple conditions. T2D requires annual reviews of 9 diabetes care processes and for patients to adopt multiple self-care tasks to prevent diabetes complications. The 9 diabetes care processes include: 3-6 monthly blood glucose measurement (HbA1c) with appropriate targets; blood pressure measurements and targets depending on diabetes complication status; annual blood cholesterol measurement; kidney function testing with urinary albumin; kidney function testing with serum creatinine; weight check; smoking status; diabetes annual eye screening; and annual foot examination.

In the National Diabetes Audit 2016-17, people with SMI and T2D were 10% less likely to take up all 9 diabetes care processes and have worse glycaemic control as a result. Therefore the aim of this study is to determine who is receiving these care processes and to develop new care pathways/interventions that support this population.

This project is a cross-sectional study and will take place in Lambeth south London, an area with high prevalence of SMI, and therefore T2D, and deprivation. W aim to profile the entire population of people with SMI and T2D within the Hills Brook and Dales and StockWELL Primary Care Networks. The investigators will access the participants medical records and record details of their latest physical health assessment and ask them to complete 7 validated questionnaires and brief informal interview either face to face in their GP surgery or over the phone. This project has been funded by the Burdett Trust for Nursing.

DETAILED DESCRIPTION:
The practice manager at each participating GP practices will run a combined search using read codes for SMI and for type 2 diabetes on the Egton Medical Information System (EMIS) electronic patient record. This will generate a list/register of all the people who potentially meet the study inclusion criteria. Next GPs or practice staff will invite the potentially eligible to participate in the study by sending them a letter and the participant information sheet. The participant will be asked to contact the research team if they would like to participate or have any further questions. If they agree to the study they receive an information sheet and consent form and will have the opportunity to ask the research team about the study.

It is expected that the total of eligible participants will be 578 from HBD and 472 for StockWELL PCN. This is because HBD PCN have a total of 57,863 patients and StockWELL have 47,199. Type 2 diabetes prevalence for Lambeth is around 5% and there are 5253 people with diabetes from the 2 PCNs which means that based on the estimated prevalence of SMI and T2D in primary care of 20%, the total population of potentially eligible participants will be in the region of 1,000. It is anticipated that 20% of people will respond to the study invitation which would mean a total population of around 200 and depending on the time available to recruit participants and the rate at which GP practices join the study and run the searches, the investigators aim to recruit at least 120 within the study period.

This will be a population-based cross-sectional survey of the total population of people with SMI and T2D registered with HBD PCN and StockWELL PCN. The research team will carry out a case note review of identifiable electronic medical records at the clinical site, information that will be selected will include the date of both diagnoses, duration of both diagnoses and medication history after consent has been obtained. This information will be written in a pseudoanonymised case report form with an ID number replacing patient identifiers and will then be kept in a locked filling cabinet in James Clerk Maxwell Building, King's College London.

The research team will ask the participant to complete 7 validated questionnaires (Diabetes Distress Scale, International Physical Activity Scale, Quality of Life Scale, self-report Global Assessment of Functioning, Alcohol Usage Disorders Identification Test, Drug Abuse Screening Test and Empower Up). This will be done either over the phone or in person and the participants GP surgery, depending on their preference.

The GP Practice will be asked to conduct a routine physical health assessment on the participant, if they have not had one in the last 3 months. This would be part of their routine clinical care and consist of HbA1c (mmol/mol); BP (mmHg); eGFR (mL/min); cholesterol (mmol/mol); BMI (m/kg2).

The research worker will then conduct a brief interview, they will rate the severity of psychiatric symptoms using a validated rating scale and they will discuss how the participant accesses support for diabetes self-management, whether they have any experience of digital interventions and their thoughts on them and finally, preferences on where and how, they receive their diabetes support. This will be carried out either over the phone or in person, depending on the participants preference and will take about 30 minutes.

If the participant lacks capacity to consent, they will be asked to consent again in a few weeks to see whether capacity has been restored. If the participant still lacks capacity or they lose capacity during the study, the participant or clinical team will be asked to elect a personal or professional and consultee. The research team will contact them and ask if they are happy to consent on the participants behalf.

ELIGIBILITY:
Inclusion Criteria:

* All participants will need to have a diagnosis of type 2 diabetes and bipolar affective disorder or psychosis.
* Capacity to consent; if participant does not currently have capacity to consent, we will ask them again in a few weeks to see whether capacity has been restored. If the participant still lacks capacity, we will ask the potential participant/their clinical team if there is a professional or a personal nominee to consent on their behalf.
* Participants must be 18 years or older.

Exclusion Criteria:

* Adults without an SMI diagnosis.
* Adults with SMI and other types of diabetes, e.g. type 1 diabetes or gestational diabetes (as different management).
* Pregnancy.
* Dementia.
* Organic psychosis.
* Moderate-severe learning disabilities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participant will all have type 2 diabetes and a severe mental illness. They will be recruited from two primary care networks (HBD and StockWELL), both of these are situated in Lambeth, London.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2022-05-03 (Actual); Primary Completion 2022-08-10 (Actual); Study Completion 2022-08-10 (Actual)

PRIMARY OUTCOMES:
Diabetes Distress Scale | 1 day
  To profile the current psychological and physical status of patients registered in the Hills Brook and Dales PCN and the StockWELL PCN. The Diabetes Distress Scale will be administered.
International Physical Activity Questionnaire | 1 day
  To profile the current psychological and physical status of patients registered in the Hills Brook and Dales PCN and the StockWELL PCN. The International Physical Activity Questionnaire will be administered.
Quality of Life Scale | 1 day
  To profile the current psychological and physical status of patients registered in the Hills Brook and Dales PCN and the StockWELL PCN. The Quality of Life Scale will be administered.
Global Assessment of Functioning | 1 day
  To profile the current psychological and physical status of patients registered in the Hills Brook and Dales PCN and the StockWELL PCN. The Global Assessment of Functioning scale will be administered.
Alcohol usage disorder identification test | 1 day
  To profile the current psychological and physical status of patients registered in the Hills Brook and Dales PCN and the StockWELL PCN. The Alcohol Usage Disorders Identification Test will be administered.
Drug abuse screening test | 1 day
  To profile the current psychological and physical status of patients registered in the Hills Brook and Dales PCN and the StockWELL PCN. The Drug Abuse Screening Test will be administered.
Brief psychiatric rating scale | 1 day
  To profile the current psychological and physical status of patients registered in the Hills Brook and Dales PCN and the StockWELL PCN. The Brief Psychiatric Rating Scale will be administered.
Empower up | 1 day
  To profile the current psychological and physical status of patients registered in the Hills Brook and Dales PCN and the StockWELL PCN. The Empower Up Questionnaire will be administered.

SECONDARY OUTCOMES:
Diabetes treatment | 1 day
  Investigators will use an open interview to find out where and how the participant would like their diabetes treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Kirsty Winkley, Principal Investigator — King's College London University
Locations (9):
- United Kingdom (9):
  - Herne Hill Group Practice, London
  - Knight's Hill, London
  - Brixton Hill, London
  - Northwood Group Practice, London
  - Binfield Road Practice, London
  - Springfield Medical Centre, London
  - Beckett House, London
  - Grantham Practice, London
  - Stockwell Group Practice, London

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data can be shared if requested.
Supporting Information: Study Protocol, ICF
Time Frame: Once the study is completed.
Access Criteria: Email Kirsty Winkley to request access.